CLINICAL TRIAL: NCT00005664
Title: Evaluation of Patients With Endocrine-Related Conditions
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000127; 00-CH-0127
Record Dates: First submitted 2000-05-17; First posted 2000-05-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12-05

CONDITIONS: Adrenal Insufficiency; Pituitary Neoplasm; Obesity
Keywords: Healthy Volunteers; Endocrine Related Conditions; Endocrine Dysfunction; Early Pubertal Development
MeSH Terms: conditions — Adrenal Insufficiency; Pituitary Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This study will evaluate patients with a variety of endocrine disorders in order to 1) learn more about conditions that affect the endocrine glands (glands that secrete hormones) and 2) to train physicians in endocrinology.

Patients of all ages with endocrine-related conditions may be eligible for evaluation under this protocol. Those enrolled may be required to provide blood, saliva, urine or stool samples, and to undergo ultrasound examination of the thyroid gland, ovaries or testes, adrenal glands or other parts of the body. Laboratory or X-ray studies may be done for diagnostic or treatment purposes. In some cases, patients will receive medical or surgical treatment for their disorder. Patients and family members of patients with a hereditary disorder may be asked to provide a blood sample for genetic analysis.

DETAILED DESCRIPTION:
This protocol is designed to allow inpatient and outpatient evaluation of adults with a variety of endocrine disorders for purposes of research and physician education in our accredited endocrinology training programs. The research-directed evaluations may include blood, saliva, or urine samples, or evaluation tissue that was routinely collected for clinical care. In some patients with endocrine disorders, laboratory or radiological studies will be performed to confirm a diagnosis or to aid in the management of the patient, using standard approaches in current clinical practice. In some cases, the patient will receive medical, radiation or surgical treatment for their disorder. The purpose of these evaluations or treatments to support our clinical training or research missions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patients of all ages with endocrine-related conditions will be eligible for this protocol.
* Both male and female subjects of all ethnic backgrounds are eligible.

EXCLUSION CRITERIA:

* Unstable patients and patients with severe organ failure that may affect/limit the endocrine work-up and exhaust Clinical Center and/or NICHD resources will be excluded if appropriate. Decisions will be made on a case by case basis by investigators.
* Subjects who are unable to provide informed consent will not be accrued; however, if patients have previously given consent, they will continue to be seen for ongoing clinical care. If they require medically-indicated procedures, we will follow NIH policy regarding obtaining consent from next of kin if they have not indicated a medical decision maker.
* Minor subjects will not be accrued; they will be referred to NICHD protocols or other NIDDK protocols for evaluation of eligibility.
* Prisoners will not be recruited. If a subject becomes incarcerated during the study, s/he may continue to participate so as to not compromise medical care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1588 (Actual)
Dates: Start 2000-05-22; Study Completion 2019-12-05

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Raff H, Sharma ST, Nieman LK. Physiological basis for the etiology, diagnosis, and treatment of adrenal disorders: Cushing's syndrome, adrenal insufficiency, and congenital adrenal hyperplasia. Compr Physiol. 2014 Apr;4(2):739-69. doi: 10.1002/cphy.c130035. PMID 24715566
- [Background] Sharma ST, Nieman LK. Prolonged remission after long-term treatment with steroidogenesis inhibitors in Cushing's syndrome caused by ectopic ACTH secretion. Eur J Endocrinol. 2012 Mar;166(3):531-6. doi: 10.1530/EJE-11-0949. Epub 2011 Dec 21. PMID 22190002